CLINICAL TRIAL: NCT02302755
Title: A Pilot, Open-Label Single Center Trial of TP10 in Pediatric and Adult Patients With C3 Glomerulopathy (C3G)
Brief Title: TP10 Use in Patients With C3 Glomerulopathy (C3G)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no recruitment
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Richard JH Smith, MD (Principal Investigator), University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIowa
Record Dates: First submitted 2014-11-05; First posted 2014-11-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Dense Deposit Disease
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening/ Active Treatment Arm (Experimental): Screening Period: This includes diagnosis confirmation, consent, required tests and vaccinations.
  Treatment Period: All patients will be enrolled through the University of Iowa. This study will follow a patient-specific TP10 dose-escalation scheme during the Induction Period and subsequent dose adjustments based on complement levels during the Maintenance Period
  Interventions: Drug: TP10

INTERVENTIONS:
Drug: TP10 — All patients will be enrolled through the University of Iowa. This study will follow a patient-specific dose-escalation scheme during the Induction Period and subsequent TP10 dose adjustments based on complement levels during the Maintenance Period.
  Other Names: sCR1

SUMMARY:
The purpose of this study is to evaluate the safety of repeated TP10 dosing in pediatric and adult patients with C3G and to evaluate the activity of TP10 in pediatric and adult patients with C3G, as measured by the proportion of patients with normalization of serum C3, serum C3 breakdown products, or alternative pathway (AP) complement activity.

DETAILED DESCRIPTION:
Overview of Study Design: This study is a pilot Phase I, open-label, non-randomized, single-arm, clinical trial of TP10 in 5 patients with C3G, aged 4 years or older. The study consists of a 4-week screening period followed by a 26-week treatment period. (See Schedule of Events, Table 1.) The 26-week treatment period is further divided into an Induction Period of up to 4 weeks, followed by a Maintenance Period, which allows for continued treatment to a total of 26 weeks.

Screening Period: Patients will be identified for possible enrollment in this study through a number of mechanisms, including physician or patient-self referral and participation in an on-going study of C3G in which renal pathology is reviewed to confirm the diagnosis of C3G and genetic and complement studies are performed. Patients who appear to meet eligibility criteria for this study upon initial review will be asked to contact Drs. Nester and Smith if they are interested in this study. Those patients who express interest in this study will be scheduled for a screening clinic visit at which time they will meet the study team and review the study design and requirements. A consent for study participation will be obtained. During this visit those events/tests noted on Table 1, Screening Visit, will be completed. If not already vaccinated within the time period of active coverage specified by the vaccine manufacturer, patients will be administered meningococcal, pneumococcal and haemophilus influenzae vaccines prior to study drug administration.

Treatment Period: All patients will be enrolled through the University of Iowa. This study will follow a patient-specific dose-escalation scheme during the Induction Period and subsequent dose adjustments based on complement levels during the Maintenance Period (as described under Investigational Product Dosing and Administration).

Safety Monitoring: Safety data for this trial will be reviewed by a Data Monitoring and Safety Person (DMSP) consisting of one reviewer who is otherwise independent of trial conduct, as well as study investigators. The DMSP will review safety data on a periodic basis based on the accrual rate and emergence of safety data. The DMSP will evaluate patient data with the purpose of identifying safety concerns that may require a modification of the current study protocol and will also be responsible for determining if criteria for halting of the trial are met (see below).

Study Stopping Rules: If any of the following criteria are met, further enrollment into the trial will be halted and the data reviewed with the DMSP. The trial will only be reopened after a mutually agreed plan is defined with the DMSP.

* Futility in the first three patients. Futility is defined as:

  - Failure during the Induction Period to normalize C3, C3 breakdown products or alternative pathway complement activity
* Any of the following toxicities in more than one patient:

  * Dose-limiting toxicity (DLT), defined as any Grade 3 or higher drug-related adverse event (AE)
  * Grade 3 or higher infection caused by encapsulated bacteria, not responsive to appropriate medical intervention within 24 hours
* Drug-related death Investigational Product Dosing and Administration Each TP10 administration will consist of a 60 (±5)-minute intravenous drip infusion using a 0.22 µm in-line filter and a controlled-rate infusion pump. Administered doses will range from 5 mg/kg to 30 mg/kg, as determined by patient-specific dose-escalation and adjustment. Any change in weight of more than 10% will require re-calculation of the administered dose; otherwise, dosing may be based on the baseline weight. All dosing will be bi-weekly during induction and weekly during maintenance.

To determine the effect of TP10 on complement and C3 convertase inhibition, complement studies will include measuring TP10 serum concentrations and serum levels of C3 and C3 breakdown products and assays of alternative pathway function. Testing will be done on serum and plasma samples obtained prior to and approximately 15 minutes post each TP10 dose. All complement studies will be performed at the University of Iowa. The following treatment plan will be followed for each patient. However, given the limited experience with TP10 in the treatment of C3G, as well as the breadth of complement studies that may be used to assess the impact of treatment, it is acknowledged that the treatment plan within this pilot study may not account for all potential clinical scenarios. Therefore, adjustments to dose level or frequency that fall outside of this plan may be implemented when determined clinically appropriate by the lead investigators at the University of Iowa. In such cases, the IRB will be notified of the plan for dose change.

Induction Period During the Induction Period, samples for complement studies will be analyzed at least weekly. The first two doses of the Induction Period will be 5 mg/kg. Intra-patient dose-escalation will subsequently occur weekly, in 5 or 10 mg/kg increments (as determined by the investigator, based on complement biomarker changes), up to a maximum dose of 30 mg/kg.

The Induction Period schedule will be modified when either of the following criteria are met:

* Dose escalation will discontinue when normalization of C3, C3 breakdown products AND/OR measure(s) of alternative and/or terminal pathway complement activity is achieved. Thereafter, the patient will receive one additional TP10 dose at the same dose level as the prior dose, and then transition to the Maintenance Period.
* If the dose level of 30 mg/kg is reached without normalization of C3, C3 breakdown products AND/OR measure(s) of alternative and/or terminal pathway complement activity, the patient may receive one additional dose of TP10 at 30 mg/kg.

  * If normalization of C3, C3 breakdown products AND/OR measure(s) of alternative and/or terminal pathway complement activity fails to occur, treatment will be discontinued.
  * If normalization of C3, C3 breakdown products AND/OR measure(s) of alternative and/or terminal pathway complement activity occurs, the patient will enter the Maintenance Period and follow rules for Maintenance Period dose adjustments.

In addition, study drug dosing will be discontinued if any additional criteria for discontinuation of study therapy (see below) are met.

Maintenance Period

Since it is quite possible that the dose required for maintenance may be significantly lower than that required during induction, the Maintenance Period will seek to identify the lowest dose that provides ongoing control of undesirable complement activity. The starting dose for TP10 Maintenance will be the same dose level as the last dose during the Induction Period; however, the Maintenance Period allows for dose decrease to 2 mg/kg, which is lower than the starting dose in the Induction Period. Samples for complement studies will be collected on each dosing day and analyzed at least weekly at University of Iowa during the Maintenance Period. Therefore, treatment decisions will be made at least weekly, and dose adjustments throughout the Maintenance period will be implemented as follows (see Section 8.3.2 for further details):

* If C3, C3 breakdown products AND/OR measure(s) of alternative and/or terminal pathway complement activity are normalized for two consecutive weeks, the next Maintenance dose may be decreased by 5 mg/kg (if the previous dose is 5 mg/kg, dosing will decrease to 2 mg/kg).

  o Note: The dose level MAY be maintained if deemed appropriate by the treating investigator, with consideration to factors such as biomarker evidence of neo-C3 convertase generation and overall profile of labs utilized for defining maintenance.
* If C3 levels have dropped >25% compared to entry into the Maintenance Period, C3 breakdown products are present (greater than normal), AND/OR measure(s) of alternative or terminal pathway complement activity have significantly changed (>50% worsening in value), the next Maintenance dose will be increased by 5 mg/kg up to a maximum of 30 mg/kg (if the previous dose is 2 mg/kg, dosing will increase to 5 mg/kg).
* If a patient has experienced dose reduction and subsequent dose escalation twice, further dose reductions may not be required, but can be implemented at the investigator's discretion. Otherwise, these patients may be maintained at the last dose that provided normalization of C3, C3 breakdown products AND/OR alternative and/or terminal pathway complement activity unless there are changes requiring a dose increased, as described above.
* If normalization of C3, C3 breakdown products AND/OR alternative and/or terminal pathway complement activity fails to occur despite receipt of 30 mg/kg twice weekly dosing for two weeks, the patient will be withdrawn from the study.

The Maintenance Period will be continued until either:

* The total study treatment period of 26 weeks has elapsed;
* Any additional criteria for discontinuation of study therapy (see below) are met.

Additional criteria for treatment discontinuation

At any point during the study, treatment will be discontinued for any of the following reasons:

* Decrease in renal function, defined by an increase in serum creatinine by 50% over baseline (last assessment prior to first TP10 dose), persistent for 4 weeks.
* Development of dose-limiting toxicity (DLT), defined as any Grade 3 or higher AE attributed to TP10 dosing, or any Grade 3 infection caused by encapsulated bacteria, not responsive to appropriate medical intervention within 24 hours. Patients who experience DLT but who are considered by the treating investigator to be potentially appropriate for further TP10 treatment may be retreated only after consultation with, and agreement from, the DMSP.
* The study is terminated (see early stopping rules).
* Request of the patient or the patient's legal representative.
* If, in the investigator's medical judgment, further participation would be injurious to the patient's health or wellbeing.
* Non-compliance of the patient.
* Pregnancy.
* Patient lost to follow-up.

Criteria for Evaluation Safety Evaluations:

Safety will be assessed by vital sign measurements, clinical laboratory tests, ECG (for patients ≥ 35 years of age) and routine physical examinations, including physical growth for children up to 18 years old and the incidence and severity of adverse events (graded according to CTCAE v 4.0).

Activity Evaluations:

Activity of TP10 in C3G will be assessed via complement studies (including but not limited to serum C3, serum C3 breakdown products, and alternate pathway activity), chronic kidney disease stage, renal biopsy (C3 deposition in the glomerular basement membrane), and renal function (proteinuria, serum creatinine).

Pharmacokinetic Evaluations:

Serum concentrations of TP10 will be measured concurrently with serum C3, C3 breakdown products, and alternative pathway complement activity in samples taken immediately before and approximately 15 minutes after TP10 infusion. No pharmacokinetic parameters will be determined in this study.

Immunological Evaluations:

Patients will be monitored for the development of antibodies to TP10.

Pharmacodynamic Evaluations:

Pharmacodynamics of TP10 will be assayed by changes in serum C3, serum C3 breakdown products and alternative pathway complement activity.

Pharmacogenomic Evaluations:

Patients will undergo genetic testing of CFH, C3, CFB and CFHR5; assays for C3Nef activity; and screening for factor H autoantibodies (FHAA) and factor B autoantibodies (FBAA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have C3G as confirmed by renal biopsy within six months of enrollment (confirmation by University of Iowa investigators is required). If the patient is post transplant, the repeat renal transplant biopsy must show C3 dominant glomerulonephritis, and the patient must have a history of known C3G in the native kidney.
2. C3 serum must be less than 75% of the lower limit of normal.
3. Signs of alternative pathway dysregulation must be present. C3 breakdown products or C3Nef activity must be detectable in plasma using assays described and validated at the University of Iowa
4. Serum creatinine level must be abnormal (>97 percentile for age or <80 ml/min using the Cockroft Gault equation for adults).
5. Must have either 24 hour urine protein >1000 mg/day, or urine protein:creatinine ratio >1.0.
6. Screening laboratory values must meet the following criteria:

   * hemoglobin ≥ 9.0 g/dL
   * platelet count ≥ 100,000/mm3
   * alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 x ULN
7. Must use adequate birth control measures.
8. Patient must be willing and able to comply with study procedures including vaccination against meningitis, haemophilus and pneumococci at least 2 weeks prior to starting the Induction Period and agree to a renal biopsy at the conclusion of the study.
9. Any anti-proteinuric medications (eg, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers) must be at a stable dose for at least four weeks prior to first dose of TP10.

Exclusion Criteria:

1. Dialysis or patients with an estimated glomerular filtration rate (eGFR; using Cockroft Gault equation) of less than 30 ml/min/1.73 m2 for over a four-week period prior to the Screening Period
2. Presence or suspicion of active or untreated systemic bacterial infection that in the opinion of the investigator precludes treatment with TP10
3. Pregnancy or lactation
4. Rituximab therapy, unless discontinued with B cell levels and immunoglobulin levels normalized by study entry
5. Patients receiving immunosuppressive therapies (except for low dose steroids [≤10 mg of prednisone or equivalent per day] given for non-C3G related conditions such as asthma). Patients receiving steroids for C3G must complete a taper prior to study entry. Exceptions will be made for renal transplant patients, who may receive any appropriate therapies as needed to maintain the transplant (i.e., to prevent rejection).
6. Receipt of any complement inhibitor within 2 months of study entry
7. Receipt of any other investigational drug or device or experimental procedures beginning four weeks prior to study enrollment
8. For renal transplant patients only: histology findings of treatable rejection (i.e. that the usual transplant physician would seek to treat). Chronic allograft nephropathy is not exclusionary provided the patient's GFR meets other entry criteria.
9. A preexisting condition with a reported association as a potential cause of C3G (i.e., Monoclonal Gammopathy of Undetermined Significance [MGUS]) or an alternate glomerular disease that may interfere with the interpretation of study results
10. Malignancy except for adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or other cancer from which the patient has been disease-free for ≥ 5 years
11. Patients with myocardial infarction (MI) within 1 year of screening, congestive heart failure, arrhythmia persistent on medication at screening or clinically evident chronic lung disease
12. Known Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C infection
13. Any medical or psychological condition that, in the opinion of the investigator, would increase the patient's risk by participation in this study or would interfere with interpretation of the study

    -

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
C3 serum measurements, serum C3 breakdown products, and/or alternative pathway (AP) complement activity. | 2 years

SECONDARY OUTCOMES:
Appropriate dose range and regimen for TP10. | 2 years
  This will be based on biologic parameters including serum levels of C3 and C3 breakdown products, assays of alternative pathway activity, and dose-limiting toxicities.

OTHER OUTCOMES:
Immunogenicity of repeat TP10 administration. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard JH Smith, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States